CLINICAL TRIAL: NCT01601236
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Adaptive Design Pilot Safety and Efficacy Study of H.P. Acthar Gel (Acthar) in Patients With Diabetic Nephropathy and Proteinuria.
Brief Title: Acthar for Treatment of Proteinuria in Diabetic Nephropathy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QSC01-DN-01
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2017-07

CONDITIONS: Diabetic Nephropathy
Keywords: H.P. Acthar Gel; Acthar; diabetic nephropathy; proteinuria; nephrotic syndrome
MeSH Terms: conditions — Diabetic Nephropathies; Proteinuria; Nephrotic Syndrome | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Intervention Model Description: The 32U group was discontinued after 2 patients met pre-specified criteria related to tolerability and patients assigned to the 32U were re-assigned to the 16U group.
Who Masked: Participant, Investigator

ARMS (6):
- Acthar 8 U (0.1 mL) daily (Experimental): Repository Corticotropin Injection
  Interventions: Drug: Repository Corticotropin Injection
- Placebo (0.1 mL) daily (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Acthar 16 U (0.2 mL) daily (Experimental): Repository Corticotropin Injection
  Interventions: Drug: Repository Corticotropin Injection
- Placebo (0.2 mL) daily (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Acthar 32 U (0.4 mL) daily (Experimental): Repository Corticotropin Injection
  Interventions: Drug: Repository Corticotropin Injection
- Placebo (0.4 mL) daily (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Repository Corticotropin Injection — H.P. Acthar Gel (repository corticotropin injection) is administered via daily SC injection for 36 weeks in the three dose groups [8 U (0.1 mL), 16 U (0.2 mL), or 32 U (0.4 mL)].
  Other Names: H.P. Acthar Gel (repository corticotropin injection); Acthar; ACTH Gel; ACTH
  Arms: Acthar 16 U (0.2 mL) daily; Acthar 32 U (0.4 mL) daily; Acthar 8 U (0.1 mL) daily
Drug: Placebo — Placebo contains the same inactive ingredients as H.P. Acthar Gel without the active pharmaceutical ingredient (API). Placebo is administered via daily SC injection for 36 weeks in equal volumes as the Acthar comparator volumes.
  Arms: Placebo (0.1 mL) daily; Placebo (0.2 mL) daily; Placebo (0.4 mL) daily

SUMMARY:
This Phase 2A study is an adaptive design pilot study investigating the efficacy and safety of daily Acthar administration in diabetic patients with nephropathy and proteinuria. Patients with type 1 diabetes mellitus (T1DM) or T2DM who currently take insulin will be enrolled and randomized into 6 study groups and will be treated with either Acthar or Placebo for 36 weeks, followed by a 4 week dose taper, and a 12 week observation period. The study will compare three dose regimens of Acthar (8 U [0.1 mL], 16 U [0.2 mL], and 32 U [0.4 mL]) to equivalent volumes of Placebo to ensure the double-blind nature of the study.

Insulin-requiring patients are being enrolled to aid compliance with the daily SC administration of study medication and to allow for ease of blood glucose control by adjustment of current insulin therapy in the event of glycemic excursions. Routine safety measures, including glycemic control, will be monitored throughout the study. The adaptive design component of the study allows for the re-assignment of the high dose group to the mid dose group if unacceptable toxicity is noted as per study protocol in the high dose group. Efficacy will be assessed by monitoring serum creatinine, calculated eGFR, and proteinuria (via urinary protein to creatinine ratio [PCR]). Serum cortisol concentration and additional biomarkers in blood and urine will also be monitored.

ELIGIBILITY:
Inclusion Criteria (numbers 2, 3, 4, 5, 6, and 7 per protocol):

* Body mass index ≤ 45 kg/m2 at screening.
* Diagnosis of T1DM or T2DM, with HbA1c ≤ 9.0% at Visit 1A. Diagnosis of T2DM should have been made at > 30 years of age (if diabetes developed at a younger age, C-peptide level may be obtained to confirmed the diagnosis).
* Currently insulin-requiring

  * Patients on oral hypoglycemic therapy plus insulin are eligible provided that oral hypoglycemic agent(s) administered and the dosing regimen(s) of oral hypoglycemic therapy have been stable for ≥ 12 weeks prior to screening. No changes in oral hypoglycemic therapy should be planned or anticipated during the treatment period.
* Renal Target Disease Requirements:

  * The average of two eGFR values collected during screening (Visits 1 and 1A) must be between 20-60 mL/min/1.73m2 (calculated using the abbreviated Modification of Diet in Renal Disease [MDRD] equation AND
  * Protein to creatinine ratio (PCR) ≥ 3.0 g/g OR total urine protein ≥ 3.0 g from the 24-hour urine collection returned at Visit 1A.
* Antihypertensive Therapy:

  * Treatment with an ACEI and/or an ARB for at least 6 weeks prior to screening Visit 1A, with stable maintenance dose for ≥ 14 days prior to screening Visit 1A. No change in ACEI or ARB therapy should be planned or anticipated for the period of the study.
  * If treated with additional antihypertensive therapy(ies), duration of therapy ≥ 30 days prior to screening Visit 1A, with stable maintenance dose for ≥ 14 days prior to screening Visit 1A.
  * If the patient has documented intolerance to ACEI and/or ARB therapy (e.g. angioedema, hyperkalemia), they may be eligible for study entry, but the Medical Monitor must be consulted in these cases prior to randomization.
* Mean systolic blood pressure ≤ 140 mmHg and diastolic blood pressure ≤ 90 mmHg on ≥ 3 seated readings taken at least 5 minutes apart during the screening period at Visit 1A.

Exclusion Criteria (numbers 2, 3, 4, 5, 7, and 11 per protocol):

* Therapies and/or Medications:

  * History of prior sensitivity to Acthar or other porcine protein products.
  * Chronic systemic corticosteroid use, defined as ≥ 20 mg of prednisone or equivalent systemic corticosteroid taken for more than 4 consecutive weeks within 6 months prior to randomization. Topical, inhaled, or intra-articular corticosteroids are allowed.
  * Planned treatment with live or live attenuated vaccines once enrolled in the study.
  * Previous treatment on a drug being investigated for the treatment of diabetic nephropathy within 6 months prior to randomization.
* Contraindication to Acthar per Prescribing Information Section 4: scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of peptic ulcer, congestive heart failure, uncontrolled hypertension, primary adrenocortical insufficiency, or adrenal cortical hyperfunction.

  * For the purpose of this study, history of peptic ulcer is defined as ≤ 6 months prior to Visit 1A.
* Diabetes Target Disease Exceptions:

  * Severely uncontrolled diabetes mellitus as judged by the Principal Investigator
  * HbA1c > 9% at screening Visit 1A.
  * Fasting serum glucose > 230 mg/dL at BOTH screening Visits 1 and 1A.
  * History of diabetic ketoacidosis or non-ketotic hyperosmolar coma within 6 months of screening.
  * History of ocular laser photocoagulation therapy within 6 months of screening OR diabetic retinopathy, diabetic macular edema, or cataracts associated with impairment of visual acuity that will affect adherence with the dosing or administration of SC injections.
  * Patients unwilling to titrate insulin for blood glucose control if adjustment of hypoglycemic therapy is required during the study.
* Renal Target Disease Exceptions:

  * History of clinical or renal biopsy evidence of non-diabetic renal disease
  * Patients requiring diagnostic or interventional procedure requiring an intravenous contrast agent must delay screening/randomization for at least 14 days
* Tuberculosis: Any patient with a positive Interferon-gamma release assay, OR signs and symptoms concerning for active tuberculosis.
* Cardiovascular:

  * History of congestive heart failure (NYHA Functional Class III-IV).
  * History of dilated cardiomyopathy with ejection fraction < 40%.

    1. Exceptions require approval by the Medical Monitor.
  * Patient has had any of the following within 3 months of screening:

    1. Unstable angina
    2. Myocardial infarction
    3. Coronary artery bypass graft or percutaneous transluminal coronary angioplasty
    4. Transient ischemic attack or cerebrovascular accident
    5. Unstable arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Questcor Investigational Site, Roseville, California
  - Questcor Investigational Site, Cooper City, Florida
  - Questcor Investigational Site, Miami Springs, Florida
  - Questcor Investigational Site, The Bronx, New York
  - Questcor Investigational Site, Columbus, Ohio
  - Questcor Investigational Site, Bethlehem, Pennsylvania
  - Questcor Investigational Site, Chattanooga, Tennessee
  - Questcor Investigational Site, Greenville, Texas
  - Questcor Investigational Site, Houston, Texas
  - Questcor Investigational Site, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial recruitment target was 40 subjects.
Pre-assignment Details: Adaptive design mandated closure of groups 5 & 6 with re-assignment of subjects to groups 3 & 4 if pre-defined tolerability criteria were met in 2 of first 6 patients.
Groups:
- Group 1: Acthar 8 U (0.1 mL) Daily: H.P. Acthar Gel (repository corticotropin injection) administered via daily subcutaneous (SC) injection for 36 weeks
- Group 2: Placebo (0.1 mL) Daily: Placebo: contains the same inactive ingredients as H.P. Acthar Gel without the active pharmaceutical ingredient (API)administered via daily SC injection for 36 weeks
- Group 3: Acthar 16 U (0.2 mL) Daily; Group 5: Acthar 32 U (0.4 mL) Daily: H.P. Acthar Gel (repository corticotropin injection) administered via daily SC injection for 36 weeks
- Group 4: Placebo (0.2 mL) Daily; Group 6: Placebo (0.4 mL) Daily: Placebo: contains the same inactive ingredients as H.P. Acthar Gel without the API administered via daily SC injection for 36 weeks
Period: Overall Study
Arm/Group | Group 1: Acthar 8 U (0.1 mL) Daily | Group 2: Placebo (0.1 mL) Daily | Group 3: Acthar 16 U (0.2 mL) Daily | Group 4: Placebo (0.2 mL) Daily | Group 5: Acthar 32 U (0.4 mL) Daily | Group 6: Placebo (0.4 mL) Daily
Started | 7 | 3 | 14 | 6 | 3 | 1
Completed | 2 | 2 | 8 | 4 | 0 | 0
Not Completed | 5 | 1 | 6 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Group 1: Acthar 8 U (0.1 mL) Daily; Group 3: Acthar 16 U (0.2 mL) Daily; Group 5: Acthar 32 U (0.4 mL) Daily: Repository Corticotropin Injection
  Repository Corticotropin Injection: H.P. Acthar Gel (repository corticotropin injection) is administered via daily SC injection for 36 weeks in the three dose groups [8 U (0.1 mL), 16 U (0.2 mL), or 32 U (0.4 mL)].
- Group 2: Placebo (0.1 mL) Daily; Group 4: Placebo (0.2 mL) Daily; Group 6: Placebo (0.4 mL) Daily: Placebo
  Placebo: Placebo contains the same inactive ingredients as H.P. Acthar Gel without the active pharmaceutical ingredient (API). Placebo is administered via daily SC injection for 36 weeks in equal volumes as the Acthar comparator volumes.
- Total: Total of all reporting groups
Arm/Group | Group 1: Acthar 8 U (0.1 mL) Daily | Group 2: Placebo (0.1 mL) Daily | Group 3: Acthar 16 U (0.2 mL) Daily | Group 4: Placebo (0.2 mL) Daily | Group 5: Acthar 32 U (0.4 mL) Daily | Group 6: Placebo (0.4 mL) Daily | Total
Number analyzed (Participants) | 7 | 3 | 14 | 6 | 3 | 1 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 9 | 5 | 2 | 0 | 24
  >=65 years | 1 | 1 | 5 | 1 | 1 | 1 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 9 | 1 | 1 | 0 | 15
  Male | 3 | 3 | 5 | 5 | 2 | 1 | 19
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 14 | 6 | 3 | 1 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Estimated Glomerular Filtration Rate (eGFR) at Visit 12
Description: Percent change in eGFR at Visit 12 (Week 36) compared to average baseline eGFR obtained during screening
Time Frame: Visit 12 (Week 36)
Population: This trial had an adaptive design that pre-specified the closure of the 32 U (units) (Group 5) in the event Acthar was not well tolerated at that dose. Based on tolerability, all patients initially included in the 32 U arm were combined with the 16 U arm (Group 3).
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo: Groups 2, 4, 6
- Acthar 8 Units: Group 1
- Acthar 16 Units: Groups 3, 5
Arm/Group | Placebo | Acthar 8 Units | Acthar 16 Units
Number analyzed (Participants) | 10 | 7 | 16
percent change | -24.927 (5.4198) | -20.563 (6.8126) | -17.447 (4.3473)

2. Secondary Outcome: Percent Change in eGFR at Visit 17
Description: Percent change in eGFR at Visit 17 (Week 52) compared to baseline eGFR obtained during screening
Time Frame: Visit 17 (Week 52)
Population: This trial had an adaptive design that pre-specified the closure of the 32 U arm (Group 5) in the event Acthar was not well tolerated at that dose. Based on tolerability, all patients initially included in the 32 U arm were combined with the 16 U arm (Group 3).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Acthar 8 Units | Acthar 16 Units
Number analyzed (Participants) | 8 | 6 | 10
percent change | -20.407 (6.0183) | -37.456 (7.8387) | -22.097 (5.4619)

3. Secondary Outcome: Frequency of Patients With a Doubling of Serum Creatinine, Progression to End-stage Renal Disease (ESRD), or Death
Time Frame: Visit 12 (Week 36) and Visit 17 (Week 52)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acthar 8 Units | Acthar 16 Units
Number analyzed (Participants) | 10 | 7 | 16
Participants
  Visit 12 (Week 36): Yes | 0 | 1 | 1
  Visit 12 (Week 36): No | 10 | 6 | 15
  Visit 17 (Week 52): Yes | 0 | 1 | 2
  Visit 17 (Week 52): No | 10 | 6 | 14

4. Secondary Outcome: Complete or Partial Remission of Proteinuria
Description: Proportion of patients with complete remission (PCR 0.5 g/g) or partial remission (reduction in PCR of >50% from baseline, plus PCR≤2.5 g/g but >0.5 g/g) of proteinuria at Visit 12 (Week 36) and/or at Visit 17 (Week 52)
Time Frame: Visit 12 (Week 36) and Visit 17 (Week 52)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acthar 8 Units | Acthar 16 Units
Number analyzed (Participants) | 9 | 3 | 8
Participants
  Visit 12 (Week 36): Complete remission | 0 | 0 | 1
  Visit 12 (Week 36): Partial remission | 1 | 0 | 0
  Visit 12 (Week 36): No remission | 8 | 3 | 7
  Visit 17 (Week 52): number analyzed (Participants) | 6 | 2 | 8
  Visit 17 (Week 52): Complete remission | 0 | 0 | 1
  Visit 17 (Week 52): Partial remission | 0 | 0 | 0
  Visit 17 (Week 52): No remission | 6 | 2 | 7

5. Secondary Outcome: Percent Change in eGFR Calculated Using Cystatin C
Description: Percent change in eGFR calculated using cystatin C compared to baseline obtained at Visit 2.
Time Frame: Visit 12 (Week 36) and Visit 17 (Week 52)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Acthar 8 Units | Acthar 16 Units
Number analyzed (Participants) | 9 | 3 | 8
percent change
  Visit 12 (Week 36) | -14.25 (17.155) | -11.49 (10.334) | -10.24 (22.066)
  Visit 17 (Week 52): number analyzed (Participants) | 6 | 2 | 8
  Visit 17 (Week 52) | 1.14 (21.155) | -35.90 (1.509) | -12.43 (20.522)

6. Secondary Outcome: Percent Change From Baseline in eGFR by Visit
Description: Percent change from baseline in eGFR by visit
Time Frame: Visit 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16 and 17
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Acthar 8 Units | Acthar 16 Units
Number analyzed (Participants) | 10 | 7 | 16
percent change
  Baseline to Visit 3: number analyzed (Participants) | 9 | 7 | 14
  Baseline to Visit 3 | -6.19 (16.494) | 1.82 (11.347) | 0.86 (11.659)
  Baseline to Visit 4: number analyzed (Participants) | 10 | 7 | 14
  Baseline to Visit 4 | -11.76 (14.131) | 4.39 (9.133) | -2.69 (11.252)
  Baseline to Visit 5: number analyzed (Participants) | 10 | 5 | 12
  Baseline to Visit 5 | -8.42 (14.942) | -10.11 (9.614) | -12.01 (14.395)
  Baseline to Visit 6: number analyzed (Participants) | 9 | 5 | 11
  Baseline to Visit 6 | -12.73 (8.881) | -9.36 (14.723) | -14.20 (16.300)
  Baseline to Visit 7: number analyzed (Participants) | 9 | 5 | 11
  Baseline to Visit 7 | -12.30 (6.888) | -25.42 (10.079) | -17.33 (21.629)
  Baseline to Visit 8: number analyzed (Participants) | 8 | 3 | 10
  Baseline to Visit 8 | -11.64 (6.539) | -27.46 (11.435) | -17.58 (23.071)
  Baseline to Visit 9: number analyzed (Participants) | 9 | 3 | 10
  Baseline to Visit 9 | -14.46 (8.535) | -21.04 (8.414) | -23.25 (18.344)
  Baseline to Visit 10: number analyzed (Participants) | 8 | 3 | 8
  Baseline to Visit 10 | -15.75 (10.914) | -28.73 (6.789) | -20.57 (23.747)
  Baseline to Visit 11: number analyzed (Participants) | 9 | 3 | 8
  Baseline to Visit 11 | -14.71 (12.052) | -26.13 (3.041) | -19.05 (20.996)
  Baseline to Visit 12: number analyzed (Participants) | 9 | 3 | 8
  Baseline to Visit 12 | -26.09 (11.687) | -23.54 (7.853) | -18.32 (22.929)
  Baseline to Week 36 Endpoint | -24.96 (11.581) | -20.27 (15.818) | -17.55 (19.655)
  Baseline to Visit 13: number analyzed (Participants) | 8 | 3 | 7
  Baseline to Visit 13 | -17.94 (14.297) | -29.37 (10.193) | -23.46 (25.490)
  Baseline to Visit 14: number analyzed (Participants) | 8 | 2 | 8
  Baseline to Visit 14 | -21.88 (11.695) | -33.99 (20.993) | -29.96 (18.970)
  Baseline to Visit 15: number analyzed (Participants) | 7 | 2 | 7
  Baseline to Visit 15 | -17.40 (14.334) | -38.05 (8.677) | -19.95 (18.899)
  Baseline to Visit 16: number analyzed (Participants) | 5 | 2 | 8
  Baseline to Visit 16 | -19.16 (18.686) | -40.18 (5.668) | -27.33 (16.709)
  Baseline to Visit 17: number analyzed (Participants) | 6 | 2 | 8
  Baseline to Visit 17 | -18.43 (12.893) | -42.70 (15.255) | -24.55 (22.322)
  Baseline to Week 52 Endpoint: number analyzed (Participants) | 8 | 6 | 10
  Baseline to Week 52 Endpoint | -20.69 (12.433) | -36.50 (11.573) | -22.44 (20.669)

7. Secondary Outcome: Percent Change From Baseline in Protein to Creatinine Ratio (PCR)
Description: Percent change from baseline in PCR
Time Frame: Visits 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16 and 17
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Acthar 8 Units | Acthar 16 Units
Number analyzed (Participants) | 10 | 7 | 16
percent change
  Baseline to Visit 4: number analyzed (Participants) | 9 | 6 | 14
  Baseline to Visit 4 | 0.3837 (31.26202) | 44.7508 (78.75623) | 32.5701 (71.34201)
  Baseline to Visit 5: number analyzed (Participants) | 10 | 5 | 10
  Baseline to Visit 5 | -13.6630 (25.57771) | 47.4429 (54.03221) | 2.0594 (59.12062)
  Baseline to Visit 6: number analyzed (Participants) | 9 | 5 | 8
  Baseline to Visit 6 | -8.3326 (36.44142) | 72.1740 (85.20350) | -1.6086 (47.69994)
  Baseline to Visit 7: number analyzed (Participants) | 9 | 5 | 9
  Baseline to Visit 7 | 2.4621 (43.42213) | 55.9950 (42.92855) | -10.6879 (50.13402)
  Baseline to Visit 8: number analyzed (Participants) | 8 | 3 | 10
  Baseline to Visit 8 | 12.6601 (51.03925) | 53.2134 (43.68087) | -8.5381 (65.06657)
  Baseline to Visit 9: number analyzed (Participants) | 9 | 3 | 9
  Baseline to Visit 9 | 27.1483 (60.72960) | 82.7319 (67.83831) | 3.6409 (54.51979)
  Baseline to Visit 10: number analyzed (Participants) | 8 | 1 | 7
  Baseline to Visit 10 | 8.2594 (45.36335) | 18.9898 | -6.7500 (64.47765)
  Baseline to Visit 11: number analyzed (Participants) | 8 | 3 | 7
  Baseline to Visit 11 | 15.1205 (92.21718) | 69.8646 (63.88789) | 0.4566 (71.78576)
  Baseline to Visit 12: number analyzed (Participants) | 9 | 3 | 8
  Baseline to Visit 12 | 21.3540 (98.45289) | 59.8357 (55.64981) | 14.4619 (66.58000)
  Baseline to Week 36 Endpoint | 19.1847 (93.07542) | 34.8848 (25.06961) | 50.2732 (85.87435)
  Baseline to Visit 14: number analyzed (Participants) | 8 | 2 | 8
  Baseline to Visit 14 | 1.1894 (44.40008) | 11.7663 (5.63288) | -16.4956 (52.71778)
  Baseline to Visit 15: number analyzed (Participants) | 7 | 2 | 7
  Baseline to Visit 15 | 0.6294 (34.89553) | 4.3807 (6.70067) | 0.0091 (81.37129)
  Baseline to Visit 16: number analyzed (Participants) | 6 | 1 | 8
  Baseline to Visit 16 | 0.0025 (47.25812) | 21.7536 | 3.6555 (74.40718)
  Baseline to Visit 17: number analyzed (Participants) | 6 | 2 | 8
  Baseline to Visit 17 | 20.8644 (88.18113) | 19.1625 (40.46023) | -6.2356 (72.81798)
  Baseline to Week 52 Endpoint: number analyzed (Participants) | 8 | 6 | 9
  Baseline to Week 52 Endpoint | 32.9735 (78.62621) | 66.7698 (84.63637) | 12.1049 (87.56153)

8. Secondary Outcome: Proportion of Subjects Whose Best Response Was Complete or Partial Remission of Proteinuria
Description: Proportion of subjects whose best response was complete remission (PCR 0.5 g/g) or partial remission (reduction in PCR of >50% from baseline, plus PCR≤2.5 g/g but >0.5 g/g) of proteinuria
Time Frame: Visit 12 (Week 36) and Visit 17 (Week 52)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acthar 8 Units | Acthar 16 Units
Number analyzed (Participants) | 10 | 7 | 16
Participants
  Week 36: Complete remission | 0 | 0 | 1
  Week 36: Partial remission | 1 | 0 | 3
  Week 36: No remission | 9 | 7 | 12
  Between Week 36 and Week 52: number analyzed (Participants) | 8 | 2 | 8
  Between Week 36 and Week 52: Complete remission | 0 | 0 | 1
  Between Week 36 and Week 52: Partial remission | 0 | 0 | 2
  Between Week 36 and Week 52: No remission | 8 | 2 | 5

9. Secondary Outcome: Percent Change From Baseline of Serum Total Cholesterol, Triglycerides, LDL, HDL, Lp(a), Albumin, and Cortisol
Description: Percent change from baseline of serum total cholesterol, triglycerides, LDL, HDL, Lp(a), albumin, and cortisol
Time Frame: Visit 6, 9, 12, and 17
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Acthar 8 Units | Acthar 16 Units
Number analyzed (Participants) | 10 | 7 | 16
percent change
  Total cholesterol - Baseline to Visit 6: number analyzed (Participants) | 9 | 5 | 11
  Total cholesterol - Baseline to Visit 6 | -7.2 (8.15) | 34.1 (23.94) | 10.1 (29.82)
  Total cholesterol - Baseline to Visit 9: number analyzed (Participants) | 9 | 3 | 10
  Total cholesterol - Baseline to Visit 9 | 13.9 (22.90) | 20.3 (27.82) | 14.2 (25.95)
  Total cholesterol - Baseline to Visit 12: number analyzed (Participants) | 9 | 3 | 8
  Total cholesterol - Baseline to Visit 12 | 3.4 (22.97) | 11.1 (24.57) | 11.1 (32.58)
  Total cholesterol - Baseline to Week 36 Endpoint: number analyzed (Participants) | 10 | 5 | 16
  Total cholesterol - Baseline to Week 36 Endpoint | 3.9 (21.74) | 26.4 (28.05) | 12.9 (24.22)
  Total cholesterol - Baseline to Visit 17: number analyzed (Participants) | 6 | 2 | 8
  Total cholesterol - Baseline to Visit 17 | 6.3 (20.82) | -12.1 (1.57) | 9.6 (33.08)
  Total cholesterol - Baseline to Week 52 Endpoint: number analyzed (Participants) | 6 | 6 | 10
  Total cholesterol - Baseline to Week 52 Endpoint | 6.3 (20.82) | 26.8 (45.79) | 9.4 (30.28)
  Triglycerides - Baseline to Visit 6: number analyzed (Participants) | 9 | 5 | 11
  Triglycerides - Baseline to Visit 6 | 1.6 (32.24) | 30.0 (34.97) | 20.5 (58.06)
  Triglycerides - Baseline to Visit 9: number analyzed (Participants) | 9 | 3 | 10
  Triglycerides - Baseline to Visit 9 | 18.4 (34.74) | 7.9 (36.59) | 31.0 (65.70)
  Triglycerides - Baseline to Visit 12: number analyzed (Participants) | 9 | 3 | 8
  Triglycerides - Baseline to Visit 12 | 8.3 (40.39) | -7.1 (25.12) | 29.2 (61.09)
  Triglycerides - Baseline to Week 36 Endpoint: number analyzed (Participants) | 10 | 5 | 16
  Triglycerides - Baseline to Week 36 Endpoint | 8.9 (38.12) | 48.8 (141.71) | 19.9 (38.54)
  Triglycerides - Baseline to Visit 17: number analyzed (Participants) | 6 | 2 | 8
  Triglycerides - Baseline to Visit 17 | 22.6 (62.47) | -37.4 (18.78) | 27.7 (63.00)
  Triglycerides - Baseline to Week 52 Endpoint: number analyzed (Participants) | 6 | 6 | 10
  Triglycerides - Baseline to Week 52 Endpoint | 22.6 (62.47) | 33.5 (76.59) | 18.2 (59.15)
  LDL-C - Baseline to Visit 6: number analyzed (Participants) | 9 | 5 | 11
  LDL-C - Baseline to Visit 6 | -4.8 (28.04) | 47.4 (35.40) | 8.1 (42.39)
  LDL-C - Baseline to Visit 9: number analyzed (Participants) | 9 | 3 | 10
  LDL-C - Baseline to Visit 9 | 16.9 (33.30) | 36.1 (50.37) | 24.5 (48.65)
  LDL-C - Baseline to Visit 12: number analyzed (Participants) | 9 | 3 | 8
  LDL-C - Baseline to Visit 12 | 16.0 (45.78) | 23.2 (45.40) | 26.4 (74.60)
  LDL-C - Baseline to Week 36 Endpoint: number analyzed (Participants) | 10 | 5 | 16
  LDL-C - Baseline to Week 36 Endpoint | 15.9 (43.16) | 42.0 (48.66) | 12.4 (54.63)
  LDL-C - Baseline to Visit 17: number analyzed (Participants) | 6 | 2 | 8
  LDL-C - Baseline to Visit 17 | 7.4 (23.12) | -9.9 (12.73) | 25.9 (86.13)
  LDL-C - Baseline to Week 52 Endpoint: number analyzed (Participants) | 6 | 6 | 10
  LDL-C - Baseline to Week 52 Endpoint | 7.4 (23.12) | 43.2 (66.57) | 24.1 (76.69)
  HDL-C - Baseline to Visit 6: number analyzed (Participants) | 9 | 5 | 11
  HDL-C - Baseline to Visit 6 | -3.2 (14.03) | 11.8 (8.94) | 18.1 (35.97)
  HDL-C - Baseline to Visit 9: number analyzed (Participants) | 9 | 3 | 10
  HDL-C - Baseline to Visit 9 | 0.0 (11.52) | 9.8 (4.12) | 3.4 (11.34)
  HDL-C - Baseline to Visit 12: number analyzed (Participants) | 9 | 3 | 8
  HDL-C - Baseline to Visit 12 | 3.7 (26.98) | 11.4 (2.70) | -6.9 (13.21)
  HDL-C - Baseline to Week 36 Endpoint: number analyzed (Participants) | 10 | 5 | 16
  HDL-C - Baseline to Week 36 Endpoint | 2.8 (25.59) | 6.7 (7.83) | 19.0 (58.40)
  HDL-C - Baseline to Visit 17: number analyzed (Participants) | 6 | 2 | 8
  HDL-C - Baseline to Visit 17 | -5.0 (7.15) | 3.0 (12.26) | -9.2 (15.91)
  HDL-C - Baseline to Week 52 Endpoint: number analyzed (Participants) | 6 | 6 | 10
  HDL-C - Baseline to Week 52 Endpoint | -5.0 (7.15) | -0.2 (17.50) | -3.2 (21.37)
  Lp(a) - Baseline to Visit 6: number analyzed (Participants) | 9 | 5 | 11
  Lp(a) - Baseline to Visit 6 | -7.2 (14.30) | 35.9 (95.42) | 22.7 (41.97)
  Lp(a) - Baseline to Visit 9: number analyzed (Participants) | 9 | 3 | 10
  Lp(a) - Baseline to Visit 9 | 1.9 (20.24) | 1.2 (9.32) | 28.0 (67.60)
  Lp(a) - Baseline to Visit 12: number analyzed (Participants) | 9 | 3 | 8
  Lp(a) - Baseline to Visit 12 | 6.1 (31.56) | 23.3 (20.74) | 10.7 (41.39)
  Lp(a) - Baseline to Week 36 Endpoint: number analyzed (Participants) | 10 | 5 | 16
  Lp(a) - Baseline to Week 36 Endpoint | 7.5 (30.07) | 49.2 (85.05) | 16.9 (48.51)
  Lp(a) - Baseline to Visit 17: number analyzed (Participants) | 6 | 2 | 8
  Lp(a) - Baseline to Visit 17 | 28.5 (57.71) | 19.9 (24.25) | 21.7 (65.09)
  Lp(a) - Baseline to Week 52 Endpoint: number analyzed (Participants) | 6 | 6 | 10
  Lp(a) - Baseline to Week 52 Endpoint | 28.5 (57.71) | 55.6 (85.65) | 21.2 (58.11)
  Serum albumin - Baseline to Visit 6: number analyzed (Participants) | 9 | 5 | 11
  Serum albumin - Baseline to Visit 6 | -1.92 (4.848) | -9.79 (7.256) | -3.78 (9.721)
  Serum albumin - Baseline to Visit 9: number analyzed (Participants) | 9 | 3 | 10
  Serum albumin - Baseline to Visit 9 | -2.49 (6.685) | -7.77 (8.638) | -3.75 (10.749)
  Serum albumin - Baseline to Visit 12: number analyzed (Participants) | 9 | 3 | 8
  Serum albumin - Baseline to Visit 12 | -0.89 (6.798) | -2.67 (14.597) | -4.09 (4.507)
  Serum albumin - Baseline to Week 36 Endpoint | -1.42 (6.629) | -5.96 (10.357) | -7.23 (6.083)
  Serum albumin - Baseline to Visit 17: number analyzed (Participants) | 6 | 2 | 8
  Serum albumin - Baseline to Visit 17 | -0.22 (9.002) | 8.06 (15.119) | -2.33 (5.898)
  Serum albumin - Baseline to Week 52 Endpoint: number analyzed (Participants) | 8 | 6 | 10
  Serum albumin - Baseline to Week 52 Endpoint | -1.77 (8.822) | -6.15 (14.379) | -2.75 (6.207)
  Cortisol - Baseline to Visit 6: number analyzed (Participants) | 9 | 5 | 11
  Cortisol - Baseline to Visit 6 | -5.86 (28.676) | 45.08 (151.882) | 180.70 (237.206)
  Cortisol - Baseline to Visit 9: number analyzed (Participants) | 9 | 3 | 10
  Cortisol - Baseline to Visit 9 | -11.23 (22.791) | 14.44 (26.399) | 50.08 (135.687)
  Cortisol - Baseline to Visit 12: number analyzed (Participants) | 9 | 3 | 8
  Cortisol - Baseline to Visit 12 | -9.44 (39.280) | 17.72 (35.704) | 52.77 (97.269)
  Cortisol - Baseline to Week 36 Endpoint | -8.36 (37.189) | 63.46 (125.208) | 64.32 (187.125)
  Cortisol - Baseline to Visit 17: number analyzed (Participants) | 6 | 2 | 8
  Cortisol - Baseline to Visit 17 | -13.11 (31.825) | 84.26 (88.861) | 7.09 (24.739)
  Cortisol - Baseline to Week 52 Endpoint: number analyzed (Participants) | 8 | 6 | 10
  Cortisol - Baseline to Week 52 Endpoint | -8.53 (28.727) | 51.82 (91.328) | 30.21 (89.880)

10. Other Pre Specified Outcome: Change in Mean HbA1c
Description: Change from baseline mean HbA1c (%) to Week 36
Time Frame: Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: %HbA1c
Arm/Group | Placebo | Acthar 8 Units | Acthar 16 Units
Number analyzed (Participants) | 9 | 3 | 8
%HbA1c | -0.22 (0.694) | -0.33 (1.429) | -0.25 (0.729)

ADVERSE EVENTS:
Time Frame: Adverse event data displayed was collected during the 36 week treatment period.
Groups:
- Acthar 16 Units: Groups 3, 5; This trial had an adaptive design that pre-specified the closure of the 32 U arm (Group 5) in the event Acthar was not well tolerated at that dose. Based on tolerability, all patients initially included in the 32 U arm were combined with the 16 U arm (Group 3). Thus, Adverse Events were not collected separately for these Arms.
- Overall: Groups 1, 2, 3, 4, 5, 6
Arm/Group | Placebo | Acthar 8 Units | Acthar 16 Units | Overall
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/7 | 0/17 | 1/34
Serious Adverse Events (participants affected / at risk) | 2/10 | 1/7 | 2/17 | 5/34
Other Adverse Events (participants affected / at risk) | 10/10 | 6/7 | 14/17 | 30/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Acthar 8 Units (N=7) | Acthar 16 Units (N=17) | Overall (N=34)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Acthar 8 Units (N=7) | Acthar 16 Units (N=17) | Overall (N=34)
Oedema peripheral (General disorders) | 2 | 3 | 8 | 13
Fatigue (General disorders) | 1 | 0 | 0 | 1
Injection site bruising (General disorders) | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 0 | 1 | 1
Oedema (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 2 | 1 | 3
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 2
Renal impairment (Renal and urinary disorders) | 0 | 0 | 2 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 3
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 2
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 1
Mastitis (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Impetigo (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Viral diarrhoea (Infections and infestations) | 0 | 0 | 1 | 1
Blood creatinine phosphokinase increased (Investigations) | 1 | 0 | 2 | 3
Blood pressure increased (Investigations) | 0 | 1 | 1 | 2
Weight increased (Investigations) | 0 | 1 | 1 | 2
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 1
Albumin urine present (Investigations) | 0 | 0 | 1 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1 | 1
Blood ketone body increased (Investigations) | 0 | 0 | 1 | 1
Protein urine present (Investigations) | 0 | 0 | 1 | 1
Urine protein/creatinine ratio increased (Investigations) | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 2
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomitting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 2 | 3
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 2 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1
Post-traumatic headache (Nervous system disorders) | 0 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 1
Retinopathy (Eye disorders) | 1 | 0 | 1 | 2
Cataract (Eye disorders) | 0 | 0 | 1 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Groups 5 & 6 were closed when 2 of the 1st 4 subjects met predefined tolerability criteria. Enrollment terminated early at 34/40 subjects due to slow recruitment.16 of 34 subjects discontinued prior to collecting primary endpoint data at week 36.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A sole participant institution shall not, without Sponsor's prior written consent, independently publish or otherwise disclose any results of this multicenter study prior to a "multicenter" publication, or 12 months after completion of the study, whichever occurs first. Institution and Principal Investigator shall have the right to publish and present the results of Institution's and Principal Investigator's activities solely in accordance with the Sponsor's written provisions.